CLINICAL TRIAL: NCT02876003
Title: An Open-Label, Single-Arm, Phase II Study to Evaluate the Efficacy, Safety and CNS Exposure of G-202 in Patients With PSMA Positive Recurrent or Progressive Glioblastoma
Brief Title: Efficacy and Safety of G-202 in PSMA-Positive Glioblastoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been withdrawn prior to enrollment.
Sponsor: GenSpera, Inc. (Industry)
Collaborators: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G-202-008
Record Dates: First submitted 2016-08-18; First posted 2016-08-23 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- G-202 (Mipsagargin) (Experimental): G-202 (Mipsagargin) administered by intravenous infusion on 3 consecutive days of a 28-day cycle
  Interventions: Drug: G-202

INTERVENTIONS:
Drug: G-202 — G-202 administered by intravenous infusion (IV, in the vein) on Days 1, 2 and 3 of each 28-day cycle until progression or development of unacceptable toxicity
  Other Names: Mipsagargin

SUMMARY:
Glioblastoma (GBM) comprises about 16% of all malignancies of the nervous system and over 50% of all gliomas. Standard of care for newly-diagnosed GBM is a combination of surgical debulking followed by concurrent radiotherapy and chemotherapy with temozolomide. Efforts to improve second-line therapy in GBM have met with only marginal success and there is a large unmet medical need for new therapies. G-202 (mipsagargin) is an example of prodrug chemotherapy. It is activated by Prostate Specific Membrane Antigen (PSMA), which is expressed by some cancer cells and in the blood vessels of most solid tumors, including GBM, but not by normal cells or blood vessels in normal tissue. It is believed that activation of the prodrug G-202 will allow the drug to kill cancer cells. This study will evaluate the activity, safety and CNS exposure of G-202 in patients with PSMA-positive recurrent or progressive GMB receiving G-202 by intravenous infusion on three consecutive days of a 28-day cycle.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to participate in this study
* Histological or radiological confirmation of glioblastoma with PSMA positivity
* Recurrent or progressive GBM following at least one (1), but no more than two (2) prior regimens; one of the prior regimens must have included surgery and/or radiotherapy
* Age >/= 18 years
* Karnofsky Performance Status (KPS) ≥ 60%
* Life expectancy > 2 months
* Adequate hematologic, renal and hepatic function
* Adequate coagulation profile
* Not pregnant, nursing or planning to become pregnant; willing to use contraception

Exclusion Criteria:

* Deteriorating neurological symptoms, or need for increasing doses of corticosteroids or new onset of seizures
* Surgical resection or major surgery within 4 weeks or stereotactic biopsy within 1 week of first G-202 treatment
* Toxicity from prior therapy (excluding alopecia) that has not resolved to ≤ Grade 1 unless otherwise specified
* Investigational or cytotoxic therapy within 28 days or nitrosoureas within 42 days of the first treatment with G-202
* Currently requiring any type of full-dose anti-coagulation treatment, systemic administration of antibiotics or chronic administration of anti-viral agents.
* History or evidence of cardiac risk, including QTc interval on screening ECG >470 msec, left ventricular ejection fraction (LVEF) < 50%, clinically significant uncontrolled arrhythmias or arrhythmia requiring treatment with the exceptions of atrial fibrillation and paroxysmal supraventricular tachycardia, history of acute coronary syndromes within 6 months prior to the first dose of study therapy (including myocardial infarction and unstable angina, coronary artery bypass graft, angioplasty, or stenting)
* Uncontrolled cardiac or coronary artery disease
* Uncontrolled hypertension (mean systolic BP ≥ 160 mm Hg and/or mean diastolic BP ≥ 100 mm Hg on 3 determinations 5 minutes apart while on 2 anti-hypertensive agents) or hypertension requiring treatment with more than 2 anti-hypertensive agents
* Severe or uncontrolled medical disease, including uncontrolled diabetes, congestive heart failure, chronic renal disease or chronic pulmonary disease
* Severe GI bleeding within 12 weeks of treatment with G-202
* Known history of HIV, hepatitis B or hepatitis C
* Documentation of keratosis follicularis (also known as Darier or Darier-White disease)
* Requirement for chronic use of strong inhibitors or inducers of cytochrome (CYP3A4) iso-enzymes
* Known hypersensitivity to any study drug component including thapsigargin derivatives, polysorbate 20, or propylene glycol
* Any other condition, including concurrent medical condition, social circumstance or drug dependency, which in the opinion of the investigator could compromise patient safety and/or compliance with study requirements
* Another primary malignancy that has not been in remission for at least 2 years; non-melanoma skin cancer, intraepithelial carcinoma of the cervix, or prostate cancer with a current PSA ≤ 0.1 ng/mL is allowed-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09; Primary Completion 2019-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
6-month progression-free survival | 6 months
  Percentage of patients who received at least 2 cycles of G-202 and have not progressed, according to criteria of the Response Assessment in Neuro-Oncology Working Group (RANO), or died within 6 months of beginning treatment with G-202

SECONDARY OUTCOMES:
Safety | Every 2 weeks for approximately 1 year
  Proportion of patients experiencing treatment-emergent adverse events
Objective tumor response rate, best overall response | Every 8 weeks for approximately one year
  Response rate assessed by RANO criteria
Duration of PFS | Every 4 weeks for approximately one year
  Duration of time from the first administration of G-202 until the first documented progression or date of death, assessed up to 12 months
Overall survival | Every 4 weeks for approximately one year
  Duration of time from the first administration of G-202 until the date of death, assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Garni Barkhoudarian, M.D., Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No